CLINICAL TRIAL: NCT00426257
Title: Phase III Randomised Clinical Trial for Stage III Ovarian Carcinoma Randomising Between Secondary Debulking Surgery With or Without Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Secondary Debulking Surgery +/- Hyperthermic Intraperitoneal Chemotherapy in Stage III Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M06OVH-OVHIPEC; 2006-003466-34 (EudraCT Number); 2006-16 (Other Grant/Funding Number: Commissie Klinische Studies)
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2017-08

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; stage III; hyperthermic intraperitoneal chemotherapy; debulking surgery; HIPEC
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Secondary debulking surgery with hyperthermic intraperitoneal chemotherapy
  Interventions: Procedure: secondary debulking with intraperitoneal chemotherapy
- 2 (Active Comparator): Secondary debulking surgery
  Interventions: Procedure: Secondary debulking

INTERVENTIONS:
Procedure: Secondary debulking — Secondary debulking
  Arms: 2
Procedure: secondary debulking with intraperitoneal chemotherapy — secondary debulking with intraperitoneal chemotherapy
  Arms: 1

SUMMARY:
This study evaluates the efficacy and safety of the addition of hyperthermic intraperitoneal chemotherapy to secondary debulking surgery in stage III ovarian cancer.

DETAILED DESCRIPTION:
Rationale: Ovarian cancer is the second most common gynaecologic cancer in the Netherlands preceded by endometrial cancer. It is however the leading cause of death among women with gynaecologic malignancies with an annual mortality rate of 9 per 100.000. The majority of the patients are diagnosed with a high stage ovarian carcinoma due to the fact that symptoms occur at a late stage of the disease and screening methods for ovarian cancer are suboptimal. Optimal treatment consists of a combination of chemotherapy and debulking surgery. Despite the appearance of localized disease and the absence of obvious residual tumour following primary treatment, the majority of patients (80%) will have persistent disease or will develop recurrent disease. Additional strategies are warranted to reduce the recurrence rate and increase disease free survival and overall survival in this group of patients.

The concept of administering intraperitoneal chemotherapy is based on the ideas on peritoneal dialysis. Intraperitoneal drug therapy is designed to maximize drug delivery to the tumour with generally acceptable systemic side effects associated with IV administration of the drug. This strategy is especially attractive for treatment of ovarian carcinoma, which remains largely restricted to the abdominal cavity for most of its natural history. So far 3 randomised controlled trials have shown an overall and progression-free survival benefit when cisplatin is administered postoperatively by the IP route in patients with stage III, optimally resected disease. These studies however found that the majority of patients did not complete all planned 6 cycles due to catheter related problems. An alternative way of administering chemotherapy intra abdominally whilst bypassing the use of a catheter intra- abdominally is provided by perfusion of the abdomen during surgery under hyperthermic conditions. This study compares the interval debulking plus or minus the perfusion of the abdomen with chemotherapy under hyperthermic conditions during surgery (OVHIPEC).

Objective: The primary objectives of this study are comparing the duration of recurrence free survival following completion of treatment between the 2 study arms.

Secondary objectives of this study involve toxicity and morbidity, quality of life, tumour response following treatment and overall survival of the study arm compared to the standard arm.

Study design: Phase III randomised trial Study population: Patients diagnosed with stage III ovarian carcinoma, peritoneal cell carcinoma or tuba carcinoma who are eligible for interval debulking surgery either following primary chemotherapy or following incomplete primary debulking and chemotherapy. Age between 18 - 76 yr old.

Intervention: One group undergoes interval debulking with hyperthermic perfusion of the abdominal cavity with cisplatin 100 mg/m2 at the end of surgery. The other group is treated by interval debulking only.

Main study parameters/endpoints: Recurrence free survival Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants of the study will be asked to fill in quality of life questionnaires (12 times in 2 year). Blood samples will be taken following written informed consent before treatment, during surgery and during follow-up visits for marker studies and proteomics studies (10 times during 2 year). For patients participating in the pharmacokinetic studies (20) 2 tissue samples will be taken from the abdominal cavity during surgery and blood samples will be taken 6 times during and after surgery.

During follow-up 3 monthly visits will be scheduled in the first 2 years and 6-monthly visits during year 3-5. During these follow-up visits routine physical exam including pelvic exam and vaginal ultrasound (optional) is performed. CT-scans will be performed in the first 2 years before randomisation and 4 times at follow-up.

Risks of participating in this trial are related to the abdominal perfusion of cisplatin. This can cause systemic effects such as: nephrotoxicity, bone marrow toxicity, neurotoxicity, and longer hospital stay. It can also increase the chance on bowel perforation of a bowel anastomoses resulting in a longer hospital stay and possibly surgical intervention. To prevent systemic side effects of intra-abdominally administered cisplatin, sodium thiosulphate is administered intravenously during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 76 years
* Histological or cytological proven primary epithelial ovarian carcinoma or peritoneal cancer (PPSC) or fallopian tube carcinoma FIGO stage III, including serous papillary adenocarcinoma, mucinous adenocarcinoma and endometrioid adenocarcinoma.
* In case of pleural effusion cytology should be negative for tumour cells
* In case diagnosis is made based on cytology only (i.e. patients treated by primary chemotherapy) additional criteria apply:

  * Normal mammogram (< 6 weeks before first registration) and
  * Presence of pelvic mass and
  * CA 125 > 200 kU/l and
  * Serum CA125/CEA ratio > 25. If the serum CA125/CEA ratio is < 25, a barium enema or colonoscopy and gastroscopy or radiological examination of the stomach should be negative for the presence of a primary tumour of the digeste tract (< 6 weeks before registration) and
  * Omental cake or other metastases larger than 2 cm in the upper abdomen and/or regional lymph node metastasis irrespective of size (CT/MRI or ultrasound or laparoscopy)
* Patients eligible for interval debulking for the following 2 reasons:

  * Primary debulking surgery not feasible due to tumour extension or general condition (patients treated by primary chemotherapy) or
  * Incomplete primary debulking with residual disease > 1 cm
* In case of primary chemotherapy:

  * Chemotherapy consists of 3 courses of carboplatin or cisplatin combined with taxol
  * Following 2 cycles of chemotherapy at least a 30% decrease in the sum of largest diameter (LD) of target lesions taking as reference the baseline sum LD (RECIST criteria, see appendix 1)
* In case of an incomplete primary debulking as indicated under 5 followed by chemotherapy:

  * Chemotherapy consists of 3 courses of carboplatin or cisplatin combined with taxol
* General criteria:

  * Fit for major surgery, ASA 1 or ASA 2
  * WHO performance status 0-2
  * Written informed consent
  * Laboratory values: serum creatinine < 140 µmol/L; creatinine clearance > 60 ml/min (Cockroft formula); white blood cell count > 3.5 x 109/l; platelets > 100 x 109 /l
* For quality of life studies:

  * Baseline questionnaires should be filled in before randomization

Exclusion Criteria:

* History of breast cancer or previous malignancies within 5 years prior to inclusion, with the exception of radically excised basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

Ages: 18 Years to 76 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2007-02; Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Duration of recurrence free survival.

SECONDARY OUTCOMES:
Toxicity and morbidity
Quality of life
Tumour response
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Willemien J van Driel, MD, Study Chair — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Derived] Aronson SL, Walker C, Thijssen B, van de Vijver KK, Horlings HM, Sanders J, Alkemade M, Koole SN, Lopez-Yurda M, Lok CAR; OVHIPEC-1 Study Group; Rottenberg S, van Rheenen J, Sonke GS, van Driel WJ, Kester LA, Hahn K. Tumour microenvironment characterisation to stratify patients for hyperthermic intraperitoneal chemotherapy in high-grade serous ovarian cancer (OVHIPEC-1). Br J Cancer. 2024 Aug;131(3):565-576. doi: 10.1038/s41416-024-02731-6. Epub 2024 Jun 12. PMID 38866963
- [Derived] Aronson SL, Lopez-Yurda M, Koole SN, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van Gent MDJM, Arts HJG, van Ham MAPC, van Dam PA, Vuylsteke P, Aalbers AGJ, Verwaal VJ, Van de Vijver KK, Aaronson NK, Sonke GS, van Driel WJ. Cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy in patients with advanced ovarian cancer (OVHIPEC-1): final survival analysis of a randomised, controlled, phase 3 trial. Lancet Oncol. 2023 Oct;24(10):1109-1118. doi: 10.1016/S1470-2045(23)00396-0. Epub 2023 Sep 11. PMID 37708912
- [Derived] Ubachs J, Koole SN, Lahaye M, Fabris C, Bruijs L, Schagen van Leeuwen J, Schreuder HWR, Hermans RH, de Hingh IH, van der Velden J, Arts HJ, van Ham M, van Dam P, Vuylsteke P, Bastings J, Kruitwagen RFPM, Lambrechts S, Olde Damink SWM, Rensen SS, Van Gorp T, Sonke GS, van Driel WJ. No influence of sarcopenia on survival of ovarian cancer patients in a prospective validation study. Gynecol Oncol. 2020 Dec;159(3):706-711. doi: 10.1016/j.ygyno.2020.09.042. Epub 2020 Oct 2. PMID 33019981
- [Derived] Koole SN, van Lieshout C, van Driel WJ, van Schagen E, Sikorska K, Kieffer JM, Schagen van Leeuwen JH, Schreuder HWR, Hermans RH, de Hingh IH, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AG, Verwaal VJ, Van de Vijver KK, Aaronson NK, van Tinteren H, Sonke GS, van Harten WH, Retel VP. Cost Effectiveness of Interval Cytoreductive Surgery With Hyperthermic Intraperitoneal Chemotherapy in Stage III Ovarian Cancer on the Basis of a Randomized Phase III Trial. J Clin Oncol. 2019 Aug 10;37(23):2041-2050. doi: 10.1200/JCO.19.00594. Epub 2019 Jun 28. PMID 31251694
- [Derived] Koole SN, Kieffer JM, K Sikorska, Schagen van Leeuwen JH, Schreuder HWR, Hermans RH, de Hingh IH, van der Velden J, Arts HJ, van Ham MAPC, Aalbers AG, Verwaal VJ, Van de Vijver KK, Sonke GS, van Driel WJ, Aaronson NK. Health-related quality of life after interval cytoreductive surgery with or without hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with stage III ovarian cancer. Eur J Surg Oncol. 2021 Jan;47(1):101-107. doi: 10.1016/j.ejso.2019.05.006. Epub 2019 May 13. PMID 31128948
- [Derived] van Driel WJ, Koole SN, Sikorska K, Schagen van Leeuwen JH, Schreuder HWR, Hermans RHM, de Hingh IHJT, van der Velden J, Arts HJ, Massuger LFAG, Aalbers AGJ, Verwaal VJ, Kieffer JM, Van de Vijver KK, van Tinteren H, Aaronson NK, Sonke GS. Hyperthermic Intraperitoneal Chemotherapy in Ovarian Cancer. N Engl J Med. 2018 Jan 18;378(3):230-240. doi: 10.1056/NEJMoa1708618. PMID 29342393